CLINICAL TRIAL: NCT02779985
Title: The Effect of a Single Dose of Lycium Barbarum on Postprandial Energy Expenditure in Healthy Overweight Men
Brief Title: Goji Berries and Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 15-3-060
Record Dates: First submitted 2016-04-18; First posted 2016-05-23 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-04

CONDITIONS: Overweight
Keywords: Lycium Barbarum; Energy expenditure; Postprandial metabolism
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lycium Barbarum mixed meal (Experimental): Subjects will receive a high-fat mixed meal containing Lycium Barbarum once.
  Interventions: Dietary Supplement: Lycium Barbarum mixed meal
- Control mixed meal (Active Comparator): Subjects will receive a high-fat mixed meal without Lycium Barbarum as a control.
  Interventions: Dietary Supplement: Control mixed meal

INTERVENTIONS:
Dietary Supplement: Lycium Barbarum mixed meal — This mixed meal contains 25 grams of dried Lycium Barbarum (Goji berry, Wolfberry)
  Arms: Lycium Barbarum mixed meal
Dietary Supplement: Control mixed meal — This mixed meal does not contain Lycium Barbarum, but is matched for energy and macronutrient content
  Arms: Control mixed meal

SUMMARY:
Effects of foods or food substances on energy expenditure are of particular interest, because of the increasing prevalence of obesity and its consequent metabolic diseases like type II diabetes and fatty liver disease, all risk factors for the development of cardiovascular diseases (CVDs). Recently, the Goji berry (Lycium Barbarum, wolfberry) was introduced into the Western diet. L. Barbarum originates from Asia, where it is used to improve the health of several organs. Although L. Barbarum is promoted as a super food with many beneficial effects, consistent scientific evidence for these effects is lacking. In one study, it was found that short-term intake of L. Barbarum polysaccharides - equal to 150 g of fresh berries - increased postprandial oxygen consumption. This indicates that L. Barbarum might exert beneficial effects on energy expenditure. Furthermore, long-term intervention trials have shown beneficial effects of L. Barbarum on lipid and glucose metabolism in mice and type II diabetic patients and on inflammatory status in healthy elderly. Altogether, L. Barbarum has the potential to be used as a functional food to increase metabolic health, but detailed information on the postprandial effects of L. Barbarum is missing. We therefore propose this double-blinded, randomized, placebo controlled intervention trial to investigate the effect of a single dose of L. Barbarum on postprandial energy expenditure substrate oxidation, metabolic flexibility, lipid and glucose metabolism and inflammatory markers.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to investigate the effect of a single dose of L. Barbarum on postprandial energy expenditure. Secondary objectives are to investigate the effect of a single dose of L. Barbarum on postprandial lipid and carbohydrate oxidation and metabolic flexibility, on postprandial lipid and glucose metabolism and on inflammatory markers.

Study design:

This is a double blind, randomized, placebo-controlled intervention trial with two test days separated by a washout period of at least 1 week.

Study population:

The study population will consist of 20 apparently healthy overweight (BMI between 25 and 30 kg/m2) men aged 18-65 years.

Intervention:

All subjects will receive a mixed meal including 25 grams of dried L. Barbarum as the intervention product and a matched mixed meal without L. Barbarum as the placebo product. The meals will be matched for energy content and macronutrient composition.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* BMI between 25 and 30 kg/m2
* Non-smoking
* Normal fasting triacylglycerol levels (<2.2 mmol/L)
* No hyperglycaemia or hypercholesterolemia (fasting glucose < 7.0 mmol/L and total cholesterol < 8.0 mmol/L)
* Willing to comply to the study protocol during the study
* Agreeing to be informed about medically relevant personal test-results

Exclusion Criteria:

* Use of anticoagulant medication
* Unstable body weight (weight gain or loss >3 kg in the past 3 months)
* Indications of treatment according to the Standard for Cardiovascular Risk Management from the Dutch General Practitioners community
* Any medical condition that might interfere with study measurements, judged by the principal investigator, including cardiovascular disease or events (e.g. acute myocardial infarction or cerebra-vascular accident), diabetes or hypercholesterolemia
* Use of any kind of medication or medically prescribed diet, which can interfere with the study (judged by the principal investigator). The use of paracetamol is allowed
* Use of oral antibiotics (with the exception of topical antibiotics) in 40 days or less prior to the start of the study
* Use of food supplements or plant-sterol/stanol-enriched foods or supplements in the three weeks prior to the screening and/or during the study
* Not willing to abstain from L. Barbarum consumption thee weeks before the start and during the trial
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, chronic obstructive pulmonary disease and rheumatoid arthritis
* Consumption of > 14 alcohol consumptions a week
* Reported intense sporting activities > 10 hours a week
* Abuse of drugs
* Participation in any other biomedical trial one month prior to the screening visit
* Having donated > 150 ml blood within 1 month prior to the screening visit, planning to donate blood during the study or within one month after finishing the study
* Impossible or difficult to puncture as evidenced during the screening visit

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline energy expenditure | Measured as the incremental area under the curve (iAUC) from 0 minutes to 140 minutes after meal intake
  Energy expenditure will be measured using indirect calorimetry (ventilated hood system). This system measures oxygen consumption (VO2) and carbon dioxide production (VCO2) to calculate the energy expenditure (kJ/min)

SECONDARY OUTCOMES:
Change from baseline energy expenditure | Measured as the incremental area under the curve (iAUC) from 160 minutes to 200 minutes and from 220 minutes to 260 minutes after meal intake
  Energy expenditure will be measured using indirect calorimetry (ventilated hood system). This system measures VO2 and VCO2 to calculate the energy expenditure (kJ/min).
Postprandial lipid and glucose oxidation | At baseline (T0, fasting) and between 0 minutes and 140 minutes, between 160 minutes and 200 minutes and between 220 minutes and 260 minutes after meal consumption
  Lipid and glucose oxidation will be calculated from indirect calorimetry data (VO2 and VCO2).
Metabolic flexibility | At 60, 120, 180 and 240 minutes after meal intake
  Metabolic flexibility will be derived from indirect calorimetry as the difference in respiratory quotient (RQ) between fasting and postprandial conditions.
Markers for lipid metabolism | At baseline (T0) and at regular intervals up to 240 minutes after meal consumption
  Several markers for lipid metabolism will be measured in blood samples.
Markers for glucose metabolism | At baseline (T0) and at regular intervals up to 240 minutes after meal consumption
  Several markers for glucose metabolism will be measured in blood samples.
Inflammatory status | At baseline (T0) and at 60, 120, 180 and 240 minutes after meal consumption
  Several markers for inflammatory status will be measured in blood samples and in vitro conditions

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Mensink, Professor, Principal Investigator — Maastricht University Medical Center; Jogchum Plat, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands